CLINICAL TRIAL: NCT00170638
Title: Tuberculosis Immunity in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 03-202
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-01

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, children, infants
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to gain a better understanding of how immunity to tuberculosis (TB) is maintained in children. When children get tuberculosis, it is more likely to spread to other parts of the body than when adults get it. This study will compare the blood cells that fight TB in children to the blood cells that fight TB in adults. Children enrolled in this study will have blood drawn on 1 or 2 occasions. Adult participants will be leukapheresed, a process in which blood passes through a machine collecting specific blood cells and returning the remaining blood to the body. An estimated 260 subjects will be enrolled in this study.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the number one cause of infectious morbidity and mortality worldwide accounting for 8 million cases and 3 million deaths annually. The impact of TB on children is particularly devastating in that children are more likely than adults to develop active TB following exposure to the bacterium, M. tuberculosis (Mtb) and once infected, children are much more likely than adults to develop disseminated disease, including miliary disease, bone and joint disease, and meningitis. These clinical differences likely reflect fundamental differences of the immune system of children and adults. The first specific aim of this study is to determine if severity of disease following Mtb infection in young children is associated with TH2-type immunity; and conversely, if absence of disease following Mtb infection is associated with TH1-type immunity by comparison of the magnitude and phenotype of Mtb-specific T cell responses in children less than or equal to 10 years old with: disseminated TB including miliary disease and meningitis; localized disease as defined by disease contained in the thoracic cavity (pulmonary, pleural, and cardiac), extrapulmonary lymph nodes (lymphadenitis), gastrointestinal tract, or bone (osteomyelitis); and latent Mtb infection (LTBI) defined as individuals with a positive Tuberculin Skin Test (TST) and without radiographic or clinical evidence of active tuberculosis. The second specific aim of this study is to determine if immunologic immaturity is associated with the development of TH2-type immunity following Mtb infection, and conversely if immunologic maturity is associated with the development of TH1-type immunity following Mtb infection by characterizing the magnitude and phenotype of Mtb-specific T cell responses in individuals with: localized disease; comparing 0-1 year olds, 2-4 year olds, 5-10 year olds, and adults; and LTBI; comparing 0-1 year olds, 2-4 year olds, 5-10 year olds, and adults. The data obtained from the present study may contribute to an improved understanding of TB immunity in children, which in turn may help in the development of a more effective TB vaccine for infants and young children. The number of participants is estimated to be 260 subjects to be enrolled over the course of 5 years.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Diagnosed with latent Mtb infection (LTBI), localized tuberculosis (TB), or disseminated TB.
* Age less than or equal to 10 years.

Adults:

* Diagnosed with localized TB or LTBI.
* All individuals with LTBI will be healthy.
* Individuals with localized TB will have been treated for TB for at least 1 month.

Exclusion Criteria:

* Older children 11-17 years old.
* Children who are immunocompromised.
* Immunocompromised adults.
* Pregnant women.
* Non-English or non-Spanish speaking individuals.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 260
Dates: Start 2005-04; Study Completion 2010-04

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States